CLINICAL TRIAL: NCT00996099
Title: Feasibility Study of the Use of Continuous Glucose Monitoring Combined With Computer-based eMPC Algorithm for Tight Glucose Control in Cardiosurgical ICU
Brief Title: Continuous Glucose Monitoring Combined With Computer Algorithm for Intensive Insulin Therapy in Cardiosurgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: prof. M. Haluzik, MD, D.Sc., 3rd Department of Medicine, Charles University, Prague
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGM-eMPC
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Hyperglycemia; Cardiac Surgery
Keywords: continuous glucose monitoring; intensive insulin therapy; critically ill; cardiac surgery; hyperglycemia of critically ill
MeSH Terms: conditions — Hyperglycemia; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CGM-eMPC (Active Comparator)
  Interventions: Device: Continuous glucose monitoring system combined with enhanced model predictive control algorithm for intensive insulin treatment
- Control (Other)
  Interventions: Other: Intensive insulin therapy using standard protocol

INTERVENTIONS:
Device: Continuous glucose monitoring system combined with enhanced model predictive control algorithm for intensive insulin treatment — Glucose measured with a real-time continuous glucose monitoring system served as an input for the enhanced model predictive control algorithm adjusting insulin infusion every 15 minutes for the first 24 hours after elective cardiac surgery
  Arms: CGM-eMPC
Other: Intensive insulin therapy using standard protocol — Insulin dosage according to the standard protocol for intensive insulin delivery used at Department of Cardiothoracic Surgery, General University Hospital, Prague.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a system combining continuous glucose measurement with a computer-based algorithm for insulin delivery in patients undergoing elective cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac surgery

Exclusion Criteria:

* insulin allergy
* mental incapacity
* language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Percentage of glycemic values in the A and B zone of Clarke Error Grid Analysis (a tool for assessing the accuracy of glucose meters) | first 24 hours after cardiac surgery

SECONDARY OUTCOMES:
Entire study average glycemia level; time within, above and below the target range throughout the whole study period and after reaching the target range | first 24 hours after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martin Haluzik, Prof, D.Sc., Principal Investigator — 3rd Department of Medicine, General University Hospital, Prague
Locations (1):
- General University Hospital, Prague, Czechia